CLINICAL TRIAL: NCT05158621
Title: A Screening Study for the Selection of Patients for Clinical Studies Targeting Tumor-specific Antigens
Brief Title: A Screening Study Targeting Tumor-specific Antigens
Status: Completed | Type: Observational
Sponsor: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GO-007
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Colorectal Cancer; Stage II/III Colon Cancer
Keywords: personalized neoantigen cancer vaccine; neoantigen cancer vaccine; individualized immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — High-Throughput Nucleotide Sequencing; Histocompatibility Testing; Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Advanced/Metastatic Colorectal Cancer: Eligible patients include those with newly-diagnosed or recurrent advanced/metastatic CRC who are initiating fluoropyrimidine and oxaliplatin (FOLFOX or CAPEOX) in combination with bevacizumab. Patients will then be assessed to determine if sufficient neoantigens are identified using Gritstone's proprietary prediction algorithm, EDGE(TM), to warrant manufacturing of an individualized vaccine. Patients with sufficient neoantigens will have vaccine manufactured while receiving FOLFOX or CAPEOX/bevacizumab.
  Interventions: Procedure: blood collection for research (next generation sequencing [NGS]); Procedure: blood collection for research (HLA typing)
- Localized Colon Cancer: Eligible patients include those with high-risk Stage II or Stage III colon cancer who have MRD based on the presence of ctDNA following surgical resection. Patients with MRD will then be assessed to determine if sufficient neoantigens are identified using Gritstone's proprietary prediction algorithm, EDGE(TM), to warrant manufacturing of an individualized vaccine.
  Interventions: Procedure: blood collection for research (next generation sequencing [NGS]); Procedure: blood collection for research (HLA typing); Procedure: blood collection for research (circulating tumor DNA [ctDNA])

INTERVENTIONS:
Procedure: blood collection for research (next generation sequencing [NGS]) — participants will have whole blood collected for NGS
Procedure: blood collection for research (HLA typing) — participants will have whole blood collected for HLA typing
Procedure: blood collection for research (circulating tumor DNA [ctDNA]) — participants will have whole blood collected for ctDNA detection
  Groups: Localized Colon Cancer

SUMMARY:
The purpose of this study is to identify patients who may be eligible to participate in a separate Phase 2/3 treatment study evaluating an individualized neoantigen vaccine GRANITE for first line (1L) maintenance treatment of metastatic, microsatellite-sable colorectal cancer (MSS-CRC) sponsored by Gritstone bio. This may include the manufacturing of an individualized vaccine, which involves neoantigen prediction and generating a vaccine targeting neoantigens.

DETAILED DESCRIPTION:
The screening study can enroll multiple tumor types in multiple treatment settings for the potential inclusion in a treatment study. Patient's tumors are analyzed to determine if the patient's tumor contains sufficient mutations. This screening study is currently enrolling patients with localized colon cancer or metastatic colorectal cancer for the development of an individualized neoantigen-based cancer vaccine that requires a manufacturing period for each patient.

The process of generating an individualized neoantigen cancer vaccine involves multiple steps, including collection of patient tumor and blood specimens, performing next-generation sequencing (NGS), predicting the neoantigens to be included in the individualized vaccine, and the manufacture and release of the individualized vaccine.

Study participants will not receive any investigational treatment as part of this trial. Patients screened in this study may be able to enroll in a separate investigational treatment study sponsored by Gritstone bio, provided that the patient meets the specified eligibility criteria for that treatment study.

ELIGIBILITY:
ADVANCED/METASTATIC COLORECTAL CANCER

Inclusion Criteria:

* signed and dated ICF prior to initiation of study-specific procedures
* histologically confirmed metastatic CRC who are planned for or who have received no more than one cycle of first-line treatment in the advanced/metastatic setting with a fluoropyrimidine and oxaliplatin in combination with bevacizumab
* measurable and unresectable disease according to RECIST v1.1
* known KRAS status
* availability of FFPE tumor specimens from biopsy within the previous 12 months for sequencing and neoantigen prediction
* ≥ 12 years of age
* ECOG performance status of 0 or 1 or equivalent for patients of 12-17 years of age
* adequate organ function (further defined in protocol)

Exclusion Criteria:

* known microsatellite instability (MSI)hi disease based on institutional standard
* known tumor mutation burden <1 nonsynonymous mutations/MB
* patients with BRAF V600E mutations

LOCALIZED COLON CANCER

Inclusion Criteria:

* signed and dated ICF prior to initiation of study-specific procedures
* high-risk stage II or stage III colon cancer planned for or have completed surgical resection and have not initiated or received more than 4 weeks of adjuvant chemotherapy and be known ctDNA-positive via the Signatera assay
* availability of FFPE tumor specimens for sequencing, determination of mutations for detecting and monitoring ctDNA to identify patients with minimal residual disease, and neoantigen prediction
* ≥ 12 years of age
* ECOG performance status of 0 or 1 or equivalent for patients of 12-17 years of age
* adequate organ function (further defined in protocol)

Exclusion Criteria:

* known microsatellite instability (MSI)hi disease based on institutional standard
* known tumor mutation burden <1 nonsynonymous mutations/MB

Complete list of inclusion and exclusion criteria are listed in the clinical study protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly-diagnosed or recurrent advanced/metastatic CRC who are initiating fluoropyrimidine and oxaliplatin (FOLFOX or CAPEOX) in combination with bevacizumab. Patients will then be assessed to determine if sufficient neoantigens are identified using Gritstone's proprietary prediction algorithm, EDGE(TM), to warrant manufacturing of an individualized vaccine.
  High-risk Stage II or Stage III colon cancer who have MRD based on the presence of ctDNA following surgical resection. Patients with MRD will then be assessed to determine if sufficient neoantigens are identified using Gritstone's proprietary prediction algorithm, EDGE(TM), to warrant manufacturing of an individualized vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Primary | at study enrollment
  To identify patients with a defined tumor-specific profile (or tumor-specific characteristics, proteins, mutations) for potential inclusion in a separate clinical study that involves investigational study treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Miami Cancer Institute, Miami, Florida
  - Advanced Research, Tamarac, Florida
  - Astera Cancer Care, East Brunswick, New Jersey
  - The Christ Hospital, Cincinnati, Ohio
  - Sarah Cannon, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia